CLINICAL TRIAL: NCT01977937
Title: Pain Control in Pediatric Posterior Spine Fusion Patients: The Effect of Gabapentin on Post-operative Opioid Use and Patient Satisfaction
Brief Title: Pain Control in Pediatric Posterior Spine Fusion Patients: The Effect of Gabapentin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Elizabeth Pedigo, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00009681
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Results first posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Pain, Postoperative
Keywords: gabapentin; Analgesic Drugs; Analgesics, Nonopioid
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gabapentin (Experimental): Gabapentin 15 milligrams per kilogram will be given orally one time pre-operatively. Gabapentin will be continued at a dose of 10 milligrams per kilogram every eight hours orally starting as soon as the patient is admitted to his or her floor bed in the hospital.
  Interventions: Drug: Gabapentin 250mg/5mL NDC:59762-5025-01
- Simple Syrup (Placebo Comparator): Simple syrup compounded by the Oregon Health and Science University research pharmacy will be administered in the same volume as if the patient were receiving the Gabapentin both pre-operatively and every eight hours after the patient is admitted to his or her floor bed in the hospital.
  Interventions: Drug: Simple Syrup

INTERVENTIONS:
Drug: Gabapentin 250mg/5mL NDC:59762-5025-01
  Arms: Gabapentin
Drug: Simple Syrup
  Arms: Simple Syrup

SUMMARY:
The purpose of this study is to evaluate the patient experience when using gabapentin with other pain control medications after posterior spinal fusion surgery for scoliosis in adolescents. These results will be compared to patients who underwent the same procedure during the study period and received the same standardized pain control regimen excluding gabapentin. Effects on pain level, opioid use, and satisfaction will be measured. Opioid side effects including nausea, sedation and urinary retention (inability to empty one's bladder) will also be recorded.The null hypotheses are as follows:

1. There is no significant difference in pain control when adding gabapentin to a multimodal pain management protocol in pediatric post-operative posterior spinal fusion patients.
2. There is no significant difference in the amount of opioid medication required for pain control in pediatric post-operative posterior spinal fusion patients.

DETAILED DESCRIPTION:
Patients aged 10-19 years with idiopathic scoliosis, and classified as American Society of Anesthesiology (ASA) class I to III who intended to undergo posterior spinal fusion for deformity correction were enrolled. Prior to surgery, subjects were randomized into either the experimental or control group by the OHSU research pharmacy using an online randomization tool, which utilized block randomization upon patient enrollment to result in equal sized groups at study completion. Patients, caretakers and providers remained blinded to the group assignments.

Patients filled out the Scoliosis Research Society, SRS-22 standardized form at a pre-operative clinic appointment. Following hospital admission, patients recorded initial pain level with the Visual Analog Scale (VAS) prior to receiving standardized pre-operative medications. The VAS scale used in this study was a 10 cm line with anchors of "no pain" at the left and "worst pain imaginable" at the right; each point was measured to the nearest millimeter. In the post-operative period, nursing staff assessed patient pain using the VAS at 4-hour intervals from 06:00 until 22:00 for the duration of hospitalization for a minimum of 4 daily scores recorded per patient. After the third post-operative day, but before discharge, the parent or guardian of each subject was asked to complete an IRB-approved survey to measure parent demographics and parental satisfaction with the patient's hospitalization and pain control.

Each patient received standardized medications according to our multimodal pain protocol. Following hospital admission, patients in both groups received one 12.5 mg/kg dose of intravenous (IV) acetaminophen. Patients in the experimental group received one 15 mg/kg dose of liquid gabapentin while the control group received a placebo, formulated to match the volume, color, taste, and smell of the experimental medication. The gabapentin or placebo was prepared by the OHSU research pharmacists so that providers and investigators remained blinded to treatment assignment. Several intraoperative anesthetic medications were given to subjects in both groups including: IV ketamine at 5mcg/kg/min for 120 minutes and IV Ketorolac 0.5mg/kg up to 15mg. Intra-operative IV propofol and IV hydromorphone were titrated to desired effect.In the post-operative period, gabapentin was administered to the experimental group at 10mg/kg PO q8h, beginning at Phase II and continued through postoperative day four. The control group received equivalent volume doses of placebo at the same intervals. Post-operative medication was administered according to the following protocol for both groups: ketorolac continued at 0.5mg/kg up to 15mg IV q6h for 12 total doses. Once ketorolac doses were complete, the patient may have received Ibuprofen 10mg/kg up to 600mg PO as needed. Hydromorphone was given through patient-controlled analgesia (PCA) at a basal dose of 0.002mg/kg/hr for 24 hours and demand dose of 0.004mg/kg with an 8-minute lockout. Once basal PCA was discontinued, administration of oxycodone 0.1-0.2mg/kg PO up to 15mg PO q4h as needed supplemented the PCA demand dose. If the patient tolerated PO oxycodone without emesis, the PCA hydromorphone was discontinued after 24 hours, but a rescue dose of hydromorphone 0.002mg IV q4 was available if needed. Other as needed medications included diazepam 0.15mg/kg up to 5mg PO q6h for muscle spasms, ondansetron 0.1mg/kg up to 4mg IV q12h for nausea, and IV acetaminophen 12.5mg/kg up to 1000mg q6h. Acetaminophen 12.5mg/kg up to 650mg PO q6h hours was administered after the IV was removed. All patients received one Senokot-S tablet and Miralax 0.8 g/kg up to 17g daily for bowel regimen.

For the entire hospitalization, nursing staff monitored vital signs and assessed sedation using the standardized Pasero Opioid-induced Sedation Scale (POSS) protocols at 4-hour intervals.16 Any POSS score of 3 or greater resulted in more frequent monitoring of respiratory status and sedation level, decreased opioid dosing, and administration of naloxone as needed. All patients were routinely monitored for known adverse gabapentin drug reactions including: peripheral edema, nausea/emesis, viral disease, ataxia, dizziness, nystagmus, somnolence, hostile behavior, fatigue and fever, Stevens-Johnson syndrome, drug hypersensitivity reactions, drug induced coma/seizure, and suicidal thoughts. Any perceived adverse reaction would have resulted in the gabapentin or placebo being stopped at the clinicians' discretion

ELIGIBILITY:
Inclusion Criteria:

* Patients of age 10-19 with an American Society of Anesthesiologists patient classification of I to III undergoing surgery to correct idiopathic or neurogenic scoliosis.

Exclusion Criteria:

* Patients who require a surgical approach or technique differing from posterior spinal fusion and/or have allergies to any of the standardized or experimental study medications: acetaminophen, gabapentin, hydromorphone, ketorolac or oxycodone.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2013-11; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Halsey, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rusy LM, Hainsworth KR, Nelson TJ, Czarnecki ML, Tassone JC, Thometz JG, Lyon RM, Berens RJ, Weisman SJ. Gabapentin use in pediatric spinal fusion patients: a randomized, double-blind, controlled trial. Anesth Analg. 2010 May 1;110(5):1393-8. doi: 10.1213/ANE.0b013e3181d41dc2. PMID 20418301

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin: Gabapentin 15 milligrams per kilogram will be given orally one time pre-operatively. Gabapentin will be continued at a dose of 10 milligrams per kilogram every eight hours orally starting as soon as the patient is admitted to his or her floor bed in the hospital.
  Gabapentin
- Simple Syrup: Simple syrup compounded by the Oregon Health and Science University research pharmacy will be administered in the same volume as if the patient were receiving the Gabapentin both pre-operatively and every eight hours after the patient is admitted to his or her floor bed in the hospital.
  Simple Syrup
Period: Overall Study
Arm/Group | Gabapentin | Simple Syrup
Started | 27 | 28
Completed | 24 | 26
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Simple Syrup | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.8 (2.0) | 14.2 (2.1) | 14.5 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 5 | 7 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 24 | 26 | 50

OUTCOME MEASURES:

1. Primary Outcome: Difference in Pain Control When Adding Gabapentin to a Multimodal Pain Management Protocol in Pediatric Post-operative Posterior Spinal Fusion Patients.
Description: Patients will rate their pain using the Visual Analog Pain Scale (VAS). The VAS is a 10 cm line with anchors of "no pain" and "worst pain imaginable." Patients rate their pain by marking on the 10 cm line where they feel their pain is at the time. The mark is then measured according to where it is along the 10 cm line and reported (range is 0.0 at the "no pain end on the left up to 10.0 at the "worst pain imaginable" on the right). Lower pain scores on the VAS scale are considered a better outcome. The numbers seen in the outcome measure data table below represent an average of the total postoperative VAS scores recorded for each patient from each arm for the duration of their hospital stay.
Time Frame: five days
Measure: Mean (Standard Deviation); unit: pain score on a scale
Arm/Group | Gabapentin | Simple Syrup
Number analyzed (Participants) | 24 | 26
pain score on a scale | 2.46 (1.74) | 3.46 (1.96)
Statistical Analysis 1: Comparison: Gabapentin vs Simple Syrup; D'Agostino & Pearson normality test was used to assess for normal distribution. Experimental & control groups were assessed for significant differences in age, hospital days, & spinal levels fused using unpaired two-tailed Student's t-test. Differences in weight & BMI were assessed using unpaired Mann-Whitney rank sum test. Differences in average VAS scores on the operative day, each post-operative day, and average total daily opioid were compared using an unpaired two-tailed Student's t-test; Test type: Other — Differences in average pre-operative & total post-operative average VAS scores were compared between groups using an unpaired Mann-Whitney rank sum test. Hospitalization outcomes including number of days to transition off PCA, number of days with Foley catheter, & episodes of nausea, emesis, or POSS > 3 were compared between groups using an unpaired two-tailed Student's t-test. Statistical significance was defined as p<0.05 for all unpaired parametric and non-parametric comparisons; p = 0.07, t-test, 2 sided

2. Secondary Outcome: Opiate Usage in the Gabapentin Group Versus Control.
Description: Total the amount of Hydromorphone and Oxycodone used in milligrams per kilogram in each patient post-operatively, convert this amount to morphine equivalents, and determine if there is a significant difference between the Gabapentin versus Placebo group.
Time Frame: Five Days
Measure: Mean (Standard Deviation); unit: morphine equivalents mg per kg
Arm/Group | Gabapentin | Simple Syrup
Number analyzed (Participants) | 24 | 26
morphine equivalents mg per kg | 3.58 (1.82) | 5.33 (3.20)
Statistical Analysis 1: Comparison: Gabapentin vs Simple Syrup; Differences in the average total daily opioid were compared between groups using an unpaired two-tailed Student's t-test; Test type: Other; p = 0.02, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the time period that patients spent in the hospital during their procedure (operative day through discharge day). Average hospital stay was 4.5 days with a standard deviation of 0.7 days for the gabapentin arm and 0.9 days for the placebo arm.
Arm/Group | Gabapentin | Simple Syrup
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 1/24 | 0/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=24) | Simple Syrup (N=26)
Emesis (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/37/NCT01977937/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT01977937/Prot_SAP_001.pdf